CLINICAL TRIAL: NCT00640536
Title: The Evaluation of Subclinical Right Ventricular Dysfunction in Obstructive Sleep Apnea Patients Without Systemic and Pulmonary Arterial Hypertension Using Velocity Vector Imaging
Brief Title: Right Ventricular Function in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Prof. Dr. Saide Aytekin, T.C. Istanbul Bilim University; Florence Nightingale Hospital
Other Study IDs: AT-1974/1
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Newly diagnosed obstructive sleep apnea patients without systemic and pulmonary arterial hypertension
- 2: Age, sex and and body mass index-matched matched healthy subjects

SUMMARY:
The purpose of this study is to determine the structural and functional cardiac alterations in obstructive sleep apne (OSA) independent from systemic and pulmonary arterial hypertension and their correlation to the severity of OSA.

DETAILED DESCRIPTION:
Many risk factors for OSA, such as male gender, obesity, and increasing age are the same as for cardiovascular diseases. This fact makes it more difficult to establish a causal relationship between OSA and cardiovascular diseases. The relationship between OSA and right ventricular (RV) function is controversial. RV dysfunction may be a result of chronic intermittent hypoxia and hypercapnia during apneic episodes. It may also occur secondary to left ventricular dysfunction as a result of increased afterload and sympathetic activity which causes secondary hypertension. As systemic hypertension is one of the most accompanying and contributing factors in OSA along with obesity, we tried to compare the effects of newly diagnosed OSA on RV function with an age and body mass index- matched control group.

ELIGIBILITY:
Inclusion Criteria:

For OSA patients (group1)

* Apnea Hypopnea Index equal or more than 15
* Epworth sleepiness scale equal or more than 10
* No previous treatment for OSA

Exclusion Criteria:

* Age < 18 years
* Known hypertension, or 24-hour mean blood pressure of 135 and/or 85 mmHg or more
* Mean pulmonary artery pressure > 25 mmHg
* Diabetes mellitus
* Left ventricular ejection fraction < 60%
* Moderate to severe valvular disease
* Cardiomyopathy
* Renal failure
* Coronary artery disease
* Obstructive or restrictive lung disease demonstrated on pulmonary function test
* Connective-tissue or chronic thromboembolic disease
* Pericardial disease
* Cancer and/or other important comorbidities with an expected survival < 2 years
* Suboptimal echocardiographic images for measurements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic, obstructive sleep apnea patients
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saide Aytekin, Principal Investigator — T.C. Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology
Locations (1):
- Florence Nightingale Hospital, Istanbul, Caglayan, Turkey (Türkiye)

REFERENCES:
- [Background] Otto ME, Belohlavek M, Romero-Corral A, Gami AS, Gilman G, Svatikova A, Amin RS, Lopez-Jimenez F, Khandheria BK, Somers VK. Comparison of cardiac structural and functional changes in obese otherwise healthy adults with versus without obstructive sleep apnea. Am J Cardiol. 2007 May 1;99(9):1298-302. doi: 10.1016/j.amjcard.2006.12.052. Epub 2007 Mar 20. PMID 17478161
- [Background] Okuda N, Ito T, Emura N, Suwa M, Hayashi T, Yoneda H, Kitaura Y. Depressed myocardial contractile reserve in patients with obstructive sleep apnea assessed by tissue Doppler imaging with dobutamine stress echocardiography. Chest. 2007 Apr;131(4):1082-9. doi: 10.1378/chest.06-2444. PMID 17426213
- [Background] Tavil Y, Kanbay A, Sen N, Ulukavak Ciftci T, Abaci A, Yalcin MR, Kokturk O, Cengel A. The relationship between aortic stiffness and cardiac function in patients with obstructive sleep apnea, independently from systemic hypertension. J Am Soc Echocardiogr. 2007 Apr;20(4):366-72. doi: 10.1016/j.echo.2006.09.005. PMID 17400115
- [Background] Tavil Y, Kanbay A, Sen N, Ciftci TU, Abaci A, Yalcin MR, Kokturk O, Cengel A. Comparison of right ventricular functions by tissue Doppler imaging in patients with obstructive sleep apnea syndrome with or without hypertension. Int J Cardiovasc Imaging. 2007 Aug;23(4):469-77. doi: 10.1007/s10554-006-9168-6. Epub 2006 Oct 20. PMID 17054014